CLINICAL TRIAL: NCT01846117
Title: Once-Daily Oral Dose of BeneFlax to Healthy Older Adults
Acronym: MOD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NHPD 186153
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Oxidative Stress; Inflammation; Aging; Pain
Keywords: lignans; oxidative stress; inflammation; aging; muscle weakness; pain
MeSH Terms: conditions — Inflammation; Pain; Muscle Weakness | interventions — secoisolariciresinol diglucoside; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- secoisolariciresinol diglucoside (Active Comparator): Secoisolariciresinol diglucoside (SDG) supplementation as 1.6g/day of BeneFlax containing 600 mg SDG. 1000 IU vitamin D as standard of care.
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside, vitamin D
- Whey powder (Placebo Comparator): Natural Factors Whey Factors whey protein (unflavored). An equal volume of measured whey protein (unflavored) to the Beneflax and 1000 IU vitamin D as standard of care.
  Interventions: Dietary Supplement: secoisolariciresinol diglucoside, vitamin D

INTERVENTIONS:
Dietary Supplement: secoisolariciresinol diglucoside, vitamin D — SDG supplementation as a packet of 1.6g/day of BeneFlax containing 600 mg SDG for 24 weeks Vitamin D Natural Product Number (NPN) 80003663 WN Pharmaceuticals Natural Factors Whey Factors
  Other Names: BeneFlax Flax Lignan Extract Archer Daniels Midland,#080001.

SUMMARY:
The investigators are investigating whether the flax lignan, secoisolariciresinol diglucoside, decreases oxidative stress and inflammation. The flax seed lignan is believed to be broken down in the body to produce the health benefits of flax. Flax lignan is separated from the whole flax seed as this compound is believed to have health effects. Decreasing oxidative stress and inflammation should improve a number of the problems associated with aging. This intervention consists of 600 milligrams of the flax lignan SDG daily or an equivalent amount of whey protein.

The investigators are comparing lignan to a placebo (whey powder) to examine whether a dietary intervention (i.e. flax seed containing lignan) might decrease oxidative stress and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 60 to 80 years residing in Saskatoon.
* Able to comply with study protocol.
* Able to follow simple instructions.

Exclusion Criteria:

* Age below 60 or above 80 years at initiation of the study.
* Individuals living in long term care homes.
* Individuals at risk of hypotension or with symptomatic hypotension.
* Fasting hypoglycemia.
* Unstable diabetes, or diabetics taking insulin (note: eligible diabetic participants will undergo additional testing during the study).
* Current cancer or diagnosed with cancer in the past 2 years.
* Women with an immediate family history or personal history of breast cancer or ovarian cancer.
* Significant liver or other gastrointestinal disorder including inflammatory bowel disease. (While constipation is the most common gastrointestinal problem in the elderly, it would not be a contraindication)
* Significant kidney disorder.
* Unstable or severe cardiac disease, recent myocardial infarction or stroke (either in past 6 months or significantly affecting physical mobility).
* Unstable other medical disease including, but not limited to, pulmonary disorder, epilepsy and genitourinary disorder.
* Migraine with aura within the last year (as this is a risk factor for stroke).
* Current diagnosis of a bleeding condition, or at risk of bleeding.
* Significant immunocompromise.
* Other unstable conditions.
* Current use of hormone replacement therapy (except thyroid medication is allowed).
* Current use of warfarin, clopidogrel, ticlopidine, dipyridamole or their analogues.
* Intolerances or allergies to flax or vitamin D.
* Allergy to whey
* Surgery within the last six months.
* Participation in any other clinical trial with an investigational agent within one month prior to randomization.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety of consumption of 600 mg/day of the flax lignan secoisolariciresinol diglucoside (SDG) in older adults (60-80 y) | 24 weeks
  Adverse event occurrences will be compared descriptively between the SDG and placebo groups. Safety will be assessed at 0, 8, 16 and 24 weeks; as part of the blood collection (urea, creatinine, total bilirubin, platelets, hematocrit, haemoglobin, mean corpuscular haemoglobin, mean corpuscular volume, white blood cell count, total protein including albumin and prealbumin, total calcium, electrolytes, glucose, liver enzymes (Aspartate transaminase (AST), Alanine Aminotransferase (ALT), Alkaline phosphatase (ALP), total protein, albumin, lipids, HbA1c (for diabetic participants). Blood pressure, pulse and respiratory rate will also be monitored at these time points.

SECONDARY OUTCOMES:
Effect of SDG on blood lipids | 24 weeks
  SDG and placebo groups will be compared at 0, 8, 16 and 24 weeks for changes in nonfasting levels of cholesterol, LDL, HDL, and triglycerides.
Effect of SDG on inflammation | 24 weeks
  SDG and placebo groups will be compared at 0, 8, 16 and 24 weeks for changes in pro-inflammatory markers (Interleukin-6 (IL-6), IL-1α, IL-1β, 8-isoprostane, Tumor necrosis factor-α (TNF-α), C-reactive protein).
Effect of SDG on quality of life | 24 weeks
  SDG and placebo groups will be compared at 0, 8, 16 and 24 weeks for changes in cognitive function, pain, and physical function.
Effect of SDG supplement on blood levels of flax lignan metabolites | 24 weeks
  SDG and placebo groups will be compared at 0, 8, 16 and 24 weeks for changes in cognitive function, pain, and physical function.
Effect of SDG supplement on fecal levels of flax lignan metabolites | 24 weeks
  To further understand the pharmacology of SDG, we will analyze fecal levels of the flax cyclolinopeptides. Levels will be determined 0 and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Jones, MD, FRCPC, Principal Investigator — University of Saskatchewan; Jane Alcorn, DVD, PhD, Study Chair — University of Saskatchewan; Susan Whiting, PhD, Study Chair — University of Saskatchewan; Kerry Mansell, BSP, PharmD, Study Chair — University of Saskatchewan; Sharyle Fowler, MD, Study Chair — University of Saskatchewan; Lilian Thorpe, MD, PhD, Study Chair — University of Saskatchewan; Thomas Hadjistavropoulos, PhD, RD, Study Chair — University of Regina
Locations (1):
- Saskatoon Centre for Patient-Oriented Research, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Alcorn J, Whiting S, Viveky N, Di Y, Mansell K, Fowler S, Thorpe L, Almousa A, Cheng PC, Jones J, Billinsky J, Hadjistavropoulos T. Protocol for a 24-Week Randomized Controlled Study of Once-Daily Oral Dose of Flax Lignan to Healthy Older Adults. JMIR Res Protoc. 2017 Feb 3;6(2):e14. doi: 10.2196/resprot.6817. PMID 28159728